CLINICAL TRIAL: NCT00741988
Title: Phase II Trial of Ixabepilone and Carboplatin With or Without Bevacizumab in Patients With Previously Untreated Advanced Non-Small-Cell Lung Cancer
Brief Title: Ixabepilone and Carboplatin +/- Bevacizumab in Advanced Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 179
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Results first posted 2013-02-27 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Advanced Disease; Untreated; Ixabepilone; Carboplatin; Bevacizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ixabepilone; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Experimental): ixabepilone 30 mg/m2 and carboplatin AUC = 6 intravenously (IV) on Day 1 of one 21-day treatment cycle.
  Interventions: Drug: Ixabepilone; Drug: Carboplatin
- Cohort B (Experimental): ixabepilone 30 mg/m2, carboplatin AUC = 6 intravenously (IV), and bevacizumab 15 mg/kg on Day 1 of one 21-day treatment cycle.
  Interventions: Drug: Ixabepilone; Drug: Carboplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Ixabepilone — ixabepilone 30 mg/m2
  Other Names: Ixempra
Drug: Carboplatin — carboplatin AUC = 6 intravenously (IV) on Day 1 of one 21-day treatment cycle.
  Other Names: Paraplatin; Paraplatin-AQ
Drug: Bevacizumab — bevacizumab 15 mg/kg on Day 1 of one 21-day treatment cycle.
  Other Names: Avastin
  Arms: Cohort B

SUMMARY:
This is a multicenter, non-randomized, Phase II study of patients with previously untreated NSCLC not amenable to radiotherapy or surgical treatment. The planned enrollment for this trial is 78 patients (including a 10% rate for inevaluable patients). There will be a total of 39 patients in each cohort (Cohorts A and B).

DETAILED DESCRIPTION:
The trial will include a lead-in phase for each cohort to assess safety. In Cohort A, 10 patients will receive ixabepilone 30 mg/m2 and carboplatin AUC = 6 intravenously (IV) on Day 1 of one 21-day treatment cycle. If no unexpected toxicities occur, Cohort A will open to enrollment. Enrollment for Cohort A will be done in two stages (after the lead-in portion is completed). The first stage for Cohort A will enroll a total of 22 patients (this will include the 10 patients from the lead-in phase). If there are at least 3 responses during stage 1, enrollment for stage 2 will proceed. For stage 2 of the study, 17 additional patients will be enrolled (for a total of 39 patients in Cohort A). During stage 1 and stage 2, patients in Cohort A will receive treatment with ixabepilone 30 mg/m2 and carboplatin AUC = 6 intravenously (IV) on Day 1 of each 21-day treatment cycle. Treatment will continue until disease progression or unacceptable toxicity occurs.

After the lead-in phase for Cohort A is completed, a similar lead-in portion, also consisting of 10 patients, will be done for Cohort B. Patients in Cohort B will receive ixabepilone 30 mg/m2, carboplatin AUC = 6 intravenously (IV), and bevacizumab 15 mg/kg on Day 1 of one 21-day treatment cycle. If no unexpected toxicities occur in this group, Cohort B will open to enrollment. Enrollment for Cohort B will also be done in two stages (after the lead-in portion is completed). The first stage for Cohort B will enroll a total of 22 patients (this will include the 10 patients from the lead-in phase). If there are at least 3 responses during stage 1, enrollment for stage 2 will proceed. For stage 2 of the study, 17 additional patients will be enrolled (for a total of 39 patients in Cohort B). During stage 1 and stage 2, patients in Cohort B will receive treatment with ixabepilone 30 mg/m2, carboplatin AUC = 6 intravenously (IV), and bevacizumab 15 mg/kg on Day 1 of each 21-day treatment cycle. Treatment will continue until disease progression or unacceptable toxicity occurs.

Unexpected toxicities include any grade 4 hematologic toxicity or grade 3/4 non hematologic toxicity that does not reverse within 7 days in more than 2 patients.

Eligible patients will receive ixabepilone, carboplatin, and bevacizumab (bevacizumab will be administered to patients in Cohort B only) at 21-day intervals. Patients will be re evaluated every 6 weeks using computerized tomography (CT) scans. Response to therapy will be assigned using Response Evaluation Criteria in Solid Tumors (RECIST) (Therasse et al. 2000) (see Section 7). Patients who have objective response or stable disease will continue treatment for 6 cycles, until the time of tumor progression or intolerable treatment-related side effects. Patients in Cohort B without progressive disease will be eligible to receive bevacizumab monotherapy for 6 additional cycles, or until undue toxicity or tumor progression occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-small-cell bronchogenic carcinoma (squamous carcinoma, adenocarcinoma, or large cell carcinoma). Cytologic specimens obtained by brushings, washings, or needle aspiration of the defined lesion are acceptable. Mixed tumors with small-cell anaplastic elements are not eligible.
2. Patients who have newly diagnosed unresectable stage III or IV disease are eligible. Patients with stage III disease should be ineligible for combined modality therapy
3. Patients must not have received any prior antineoplastic chemotherapy for metastatic lung cancer prior to study entry.
4. Patients who have had previous radiotherapy as definitive therapy for locally advanced non-small-cell are eligible as long as the recurrence is outside the original radiation port. Radiation therapy must have been completed greater than 4 weeks prior to registration.
5. Male or female patients >=18 years of age.
6. Life expectancy of at least 3 months.
7. ECOG performance status of <=1.
8. Measurable disease by RECIST criteria (see Section 7).
9. Laboratory values as follows:

   * ANC >=1500/mm3 (7 days prior to treatment);
   * Hemoglobin >=8 g/dL;
   * Platelets >=100,000 mm3 (7 days prior to treatment)
   * Bilirubin <=1 x ULN for institution
   * AST/SGOT <=2.5 x ULN or <=5.0 x ULN in patients with liver metastases and
   * ALT/SGPT <=2.5 x ULN or <=5.0 x ULN in patients with liver metastases
   * Creatinine <=2.0 mg/dL or
   * Calculated (measured) GFR >=40 mL/min
   * PT/INR and PTT <=1.5 x ULN
10. Peripheral neuropathy <= grade 1.

Exclusion Criteria:

1. A history of cardiac disease as defined by malignant hypertension, unstable angina, congestive heart failure of > grade 2 per New York Heart Association (NYHA) criteria (see Appendix B), myocardial infarction within the previous 6 months, or symptomatic cardiac arrhythmias.
2. Metastatic brain or meningeal tumors.
3. Uncontrolled intercurrent illness.
4. Chemotherapy, investigational drug therapy, or major surgery ≤ 4 weeks prior to starting study drug, or patients who have not recovered from side effects of previous therapy.
5. Patient is <=5 years free of another primary malignancy, except if the other primary malignancy is not currently clinically significant or requiring active intervention, or if the other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ.

Exclusion Criteria for Enrollment on Bevacizumab (Cohort B):

1. Patients with squamous cell histology NSCLC.
2. Patients who have had a major surgical procedure (not including mediastinoscopy), open biopsy, or significant traumatic injury within 1 month of beginning bevacizumab.
3. Patients who have had primary thoracic radiation within 3 months of beginning bevacizumab.
4. Fine needle aspiration, core biopsy, mediastinoscopy or other minor surgical procedure within 7 days of beginning bevacizumab.
5. Patients receiving thrombolytic therapy within 10 days of starting bevacizumab.
6. Patients with serious non-healing wound, ulcer, or bone fracture.
7. Patients with evidence of bleeding diathesis or coagulopathy.
8. Patients with history of hemoptysis (defined as bright red blood of ½ teaspoon or more per episode) within 3 months prior to study enrollment.
9. Patients with proteinuria at screening, as demonstrated by either:

   * Urine protein : creatinine (UPC) ratio >=1.0 or
   * Urine dipstick for protein >=2+ (patients discovered to have >=2+ proteinuria on dipstick at baseline should undergo a 24-hour urine collection, and must demonstrate <1 g of protein in 24 hours to be eligible).
10. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to beginning bevacizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Spigel, MD, Study Chair — Sarah Cannon Research Insititute
Locations (13):
- United States (13):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Gainsville Hematology Oncology Associates, Gainesville, Florida
  - Providence Medical Group, Terre Haute, Indiana
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Research Medical Center, Kansas City, Missouri
  - Dr. Donald Berdeaux, Great Falls, Montana
  - Oncology Hematology Care, Cincinnati, Ohio
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Peninsula Cancer Institute, Newport News, Virginia

REFERENCES:
- [Result] Spigel DR, Anthony Greco F, Waterhouse DM, Shipley DL, Zubkus JD, Bury MJ, Webb CD, Hart LL, Gian VG, Infante JR, Burris HA 3rd, Hainsworth JD. Phase II trial of ixabepilone and carboplatin with or without bevacizumab in patients with previously untreated advanced non-small-cell lung cancer. Lung Cancer. 2012 Oct;78(1):70-5. doi: 10.1016/j.lungcan.2012.06.008. Epub 2012 Sep 1. PMID 22947511

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixabepilone/Carboplatin: ixabepilone 30 mg/m2 and carboplatin AUC = 6 intravenously (IV) on Day 1 of one 21-day treatment cycle.
- Ixabepilone/Carboplatin/Bevacizumab: ixabepilone 30 mg/m2, carboplatin AUC = 6 intravenously (IV), and bevacizumab 15 mg/kg on Day 1 of one 21-day treatment cycle.
Period: Overall Study
Arm/Group | Ixabepilone/Carboplatin | Ixabepilone/Carboplatin/Bevacizumab
Started | 42 | 40
Completed | 38 | 36
Not Completed | 4 | 4
Not completed — Adverse Event | 2 | 4
Not completed — Lack of Efficacy | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixabepilone/Carboplatin | Ixabepilone/Carboplatin/Bevacizumab | Total
Number analyzed (Participants) | 42 | 40 | 82
Age, Continuous [Median (Full Range); unit: years] | 63 [43 to 85] | 63 [45 to 78] | 63 [43 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 24 | 19 | 43
Region of Enrollment [Number; unit: participants]
  United States | 42 | 40 | 82

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR), the Percentage of Patients Who Experience an Objective Benefit From Treatment
Description: The Percentage of Patients Who Experience an Objective Benefit From Treatment
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixabepilone/Carboplatin | Ixabepilone/Carboplatin/Bevacizumab
Number analyzed (Participants) | 38 | 36
percentage of participants | 29 [16 to 45] | 50 [34 to 66]

2. Secondary Outcome: Progression Free Survival, the Length of Time, That Patients Were Alive From Their First Date of Treatment Until Worsening of Their Disease
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone/Carboplatin | Ixabepilone/Carboplatin/Bevacizumab
Number analyzed (Participants) | 42 | 40
months | 5.3 [2.8 to 8.6] | 6.7 [5.1 to 8.4]

3. Secondary Outcome: Overall Survival (OS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone/Carboplatin | Ixabepilone/Carboplatin/Bevacizumab
Number analyzed (Participants) | 42 | 40
months | 9.3 [6.4 to 16.6] | 13.2 [8.9 to NA] — Upper limit not reached due to patients remaining on treatment at time of analysis.

4. Secondary Outcome: Number of Participants Experiencing Treatment Related Toxicity
Description: Number of participants experiencing Grade 3 and Grade 4 Treatment-related toxicities are reported here. Toxicities that were occurring >=5% of total patients are listed. Toxicity was assessed using the Common Terminology Criteria for Adverse Events (CTCAE version 3.0) of the National Cancer Institute.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ixabepilone/Carboplatin | Ixabepilone/Carboplatin/Bevacizumab
Number analyzed (Participants) | 42 | 40
Participants
  Anemia | 4 | 6
  Leukopenia | 6 | 9
  Neutropenia | 13 | 19
  Febrile neutropenia | 1 | 1
  Cardiac arrhythmia | 2 | 0
  Dehydration | 3 | 3
  Diarrhea | 3 | 3
  Fatique | 4 | 9
  Hyponatremia | 2 | 1
  Infection | 2 | 8
  Pain (all types) | 4 | 11
  Dyspnea | 4 | 4
  Thrombocytopenia | 8 | 8
  Vomiting | 0 | 4
  Hemorrhagic events (all) | 0 | 1
  allergic (HSR) | 0 | 2
  Cough | 0 | 4

ADVERSE EVENTS:
Arm/Group | Ixabepilone/Carboplatin | Ixabepilone/Carboplatin/Bevacizumab
Serious Adverse Events (participants affected / at risk) | 14/42 | 18/40
Other Adverse Events (participants affected / at risk) | 42/42 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixabepilone/Carboplatin (N=42) | Ixabepilone/Carboplatin/Bevacizumab (N=40)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Allergic Reaction (Immune system disorders) | 0 (0) | 1 (1)
Cardiac Ischemia/Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Supraventricular arrhythmia - Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1) | 3 (4)
Hemorrhage, Pulmonary/Upper Respiratory - Hemoptysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Neuropathy - Motor (Nervous system disorders) | 1 (1) | 0 (0)
Infection - NOS (Infections and infestations) | 0 (0) | 2 (2)
Infection - Renal/Genitourinary (Infections and infestations) | 0 (0) | 1 (2)
Pain - Abdomen (General disorders) | 0 (0) | 2 (2)
Mental Status (Psychiatric disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Infection - Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Immune system disorders) | 1 (1) | 0 (0)
Neurology - Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary - Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wound Complication (Surgical and medical procedures) | 0 (0) | 1 (1)
Perforation, GI (Gastrointestinal disorders) | 0 (0) | 2 (2)
Neutrophils (Immune system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixabepilone/Carboplatin (N=42) | Ixabepilone/Carboplatin/Bevacizumab (N=40)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 6 (8) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 15 (52) | 16 (66)
Anorexia (Gastrointestinal disorders) | 13 (37) | 17 (62)
Constipation (Gastrointestinal disorders) | 17 (39) | 14 (46)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (30) | 15 (56)
Dehydration (Gastrointestinal disorders) | 9 (14) | 8 (12)
Diarrhea (Gastrointestinal disorders) | 12 (31) | 10 (38)
Dizziness (Nervous system disorders) | 9 (17) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (50) | 18 (56)
Edema - Limb (Blood and lymphatic system disorders) | 0 (0) | 10 (23)
Fatigue (General disorders) | 31 (125) | 30 (210)
Fever (General disorders) | 0 (0) | 8 (12)
Hemoglobin (Blood and lymphatic system disorders) | 35 (132) | 30 (172)
Hemorrhage - Urinary (Blood and lymphatic system disorders) | 0 (0) | 6 (12)
Hemorrhage - Nose (Blood and lymphatic system disorders) | 0 (0) | 10 (22)
Hypercalcemia (Metabolism and nutrition disorders) | 5 (11) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (21) | 5 (10)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (8) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 5 (16)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 5 (11) | 6 (16)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 8 (17)
Hypotension (Cardiac disorders) | 5 (17) | 0 (0)
Infection - NOS (Infections and infestations) | 14 (30) | 12 (31)
Insomnia (General disorders) | 9 (23) | 12 (31)
Leukocytes (Immune system disorders) | 26 (71) | 28 (78)
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 7 (14) | 5 (12)
Mood Alteration - Anxiety (Psychiatric disorders) | 0 (0) | 7 (25)
Mucositis/Stomatitis (Gastrointestinal disorders) | 0 (0) | 10 (28)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (18)
Nausea (Gastrointestinal disorders) | 23 (56) | 23 (64)
Neuropathy - Sensory (Nervous system disorders) | 15 (52) | 16 (91)
Neutrophils (Immune system disorders) | 29 (67) | 28 (64)
Pain (General disorders) | 28 (150) | 31 (232)
Platelets (Blood and lymphatic system disorders) | 23 (61) | 26 (83)
Proteinuria (Renal and urinary disorders) | 0 (0) | 13 (35)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (15)
Taste Alteration (Gastrointestinal disorders) | 6 (17) | 12 (50)
Supraventricular arrhythmia - Atrial fibrillation (Cardiac disorders) | 5 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 18 (32) | 16 (39)
Weight Loss (Metabolism and nutrition disorders) | 0 (0) | 11 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites